CLINICAL TRIAL: NCT02039076
Title: A Five-Treatment-Period Study to Evaluate the Single-Dose Pharmacokinetics and Pharmacodynamics of Avatrombopag in Healthy Japanese and White Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E5501-A001-018
Record Dates: First submitted 2014-01-13; First posted 2014-01-17 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-11

CONDITIONS: Thrombocytopenia
Keywords: Healthy
MeSH Terms: conditions — Thrombocytopenia | interventions — avatrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- avatrombopag (Experimental): Each subject will receive a single administration during each of the 5 treatment periods as follows: 40 and 60 mg in the fed and fasted state, and 20 mg in the fed state. Subjects will be randomized to one of four dosing sequences.
  Interventions: Drug: avatrombopag

INTERVENTIONS:
Drug: avatrombopag

SUMMARY:
This will be a randomized, open-label, 5-treatment-period study to evaluate the PK and PD of avatrombopag following a single administration of avatrombopag in the fed and fasted condition, or the fed condition, to healthy Japanese and white subjects. A standard high-fat, high calorie breakfast will be used to assess the fed condition.

DETAILED DESCRIPTION:
The study will comprise a Prerandomization Phase and a Randomization Phase. The Prerandomization Phase will include 2 periods, Screening and Baseline 1. The Screening Period will be up to 3 weeks (21 days) in duration. The Randomization Phase will consist of 5 single-dose treatment periods, of which 3 will include administration of avatrombopag in the fed condition and 2 will include administration of avatrombopag in the fasted condition. Each treatment period will be separated by a wash out interval of at least 28 days. Before each treatment period, subjects will complete a baseline period (Baseline Periods 2, 3, 4, and 5), during which baseline assessments will be collected. A Final Visit will occur 28 days (+/- 1 day) after dosing in Treatment Period 5.

ELIGIBILITY:
Inclusion Criteria

1. Platelet count between the lower limit of normal and 350 x 109/L, inclusive, at Screening and each Baseline; measurements can repeated for verification, if necessary
2. Nonsmoking, healthy white and Japanese adult male and female subjects, greater than or equal to 20 years and less than or equal to 55 years old at the time of informed consent. (Nonsmokers are defined as those who have discontinued smoking for at least 4 weeks before dosing.)
3. Japanese subjects must be born in Japan of Japanese parents and Japanese grandparents, must have lived no more than 5 years outside of Japan, and must not have changed their lifestyle or habits, including diet, while living outside of Japan.
4. Body mass index greater than or equal to 18 and less than or equal to 28 kg/m2 at Screening and Baseline Period 1. The BMI in white subjects must be within +/- 2 kg/m2 of the BMI in Japanese subjects.
5. Nonsmoking, healthy white and Japanese adult males and females between the ages of 20 and 55, inclusive
6. BMI between 18 and 28. inclusive
7. Females must not be pregnant or lactating, and if they are of childbearing potential they must agree to use a highly effective method of contraception or abstain
8. Males must have a vasectomy or they and their partner must use a highly effective method of contraception

Exclusion Criteria

1. Evidence of organ dysfunction or any clinically significant deviation from normal in their medical history (eg, history of splenectomy); history of arterial or venous thrombosis, including partial or complete thromboses (eg, stroke, transient ischemic attack, myocardial infarction, deep vein thrombosis, pulmonary embolism); known family history of hereditary thrombophilic disorders (eg, Factor V Leiden, antithrombin III deficiency)
2. Recent clinically significant illness or infection that requires medical treatment
3. Evidence of disease that may influence the outcome of the study (eg, psychiatric disorders, disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system), or subjects who have a congenital abnormality in metabolism
4. Any history of gastrointestinal surgery (eg, hepatectomy, nephrotomy, digestive organ resection)
5. Any clinically abnormal symptom or organ impairment found by medical history, physical examination, vital sign electrocardiogram (ECG) assessment, or laboratory test results
6. A known or suspected history of drug or alcohol dependency or abuse or a positive urine drug, cotinine, or alcohol test
7. Positive results for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibody at Screening
8. Weight loss or gain of >10% within 4 weeks before dosing
9. Known history of clinically significant drug or food allergy
10. Currently enrolled in another clinical trial

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2013-12; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) profiles of avatrombopag | Up to 23 Weeks
  The following PK parameters will be estimated for plasma: Cmax, AUC, and t1/2.

SECONDARY OUTCOMES:
Pharmacodynamic (PD) profiles of avatrombopag | Up to 23 Weeks
  Analyses will carried out for AUEC(0-28d) and Emax using a mixed linear model including fixed terms for dose, race, food, sequence, and period with interaction terms for food by race and for dose by race and subject as random effect.
Comparison of PK and PD for avatrombopag | Up to 23 Weeks
  To assess the similarity of the PK and PD of avatrombopag between healthy Japanese and white subjects after a single administration of avatrombopag under fasted conditions
Adverse events (AEs ) as a measure of safety and tolerability | Up to 23 Weeks
  Saftey assessments include AEs, clinical laboratory results, vital signs, and ECGs.
Laboratory assessments as a measure of safety and tolerability | Up to 23 Weeks
  Clinical laboratory assessments will include haematology, clinical chemistry, urinalysis and other screening tests
Vital signs as a measure of safety and tolerability | Up to 23 Weeks
  Vital sign measurements will include systolic and diastolic blood pressure (BP) and pulse rate
Electrocardiogram (ECG) as a measure of safety and tolerability | Up to 23 Weeks
  Twelve-lead ECGs will be obtained as a measure of safety and tolerability

CONTACTS AND LOCATIONS:
Locations (1):
- Parexel International Early Development Clinical Units, Glendale, California, United States